CLINICAL TRIAL: NCT04076280
Title: Sodium Watchers Program - Hypertension
Acronym: SWAPHTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misook L. Chung (Other)
Responsible Party: Sponsor-Investigator, Misook L. Chung, Professor College of Nursing, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44336
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Hypertension
Keywords: Hypertension; Low Sodium Diet
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SWAP Intervention (Experimental): The participants are randomized using a table of random numbers pre-generated by a computer assigning them to the Sodium Watcher Program.
  Interventions: Behavioral: Sodium Watcher Program-Hypertension
- Usual Care (Active Comparator): The participants are randomized using a table of random numbers pre-generated by a computer assigning them to the usual care group.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Sodium Watcher Program-Hypertension — The Sodium Watcher Program -Hypertension intervention consists of 14 weeks of education [4 weekly education sessions (45 minutes)followed by 5 bi-weekly sessions 5-20 minutes] that will be held at the dyads' preferred time delivered to their homes using a video conferencing program through an iPad.
  Arms: SWAP Intervention
Behavioral: Usual Care — Participants in the usual care group receive their routine medical and nursing care for hypertension that consists of a recommendation to follow a sodium restricted diet and take medications as ordered. Usual care consists of recommendations to follow a sodium restricted diet, but without explicit skills training including instructions on gradual adaptation to sodium restricted diet, follow-up of progress or provision of monitoring.
  Arms: Usual Care

SUMMARY:
Hypertensive adults are a vulnerable population at high risk of developing cardiovascular disease. Despite the many interventions tested to reduce hypertension, it remains a major risk factor that is not appropriately managed in the population. Prior dietary interventions were successful on reduction of sodium intake, but the changes were not maintained after the end of the intervention. We propose that changing patients' salt taste preference and including family members will produce long-term changes in sodium intake and blood pressure. The Sodium Watchers Program (SWaP) proposed in this study is designed to improve adherence to a sodium restricted diet through education and self-care strategies for gradual taste adaptation to low salt foods. The purpose of this pilot is to test short-term effects of the SWaP intervention on adherence to the sodium restricted diet, blood pressure, salt taste preference, and dietary patterns in hypertensive adults. A total of 30 hypertensive adults will be randomly assigned to the intervention (n=20) or control group (n=10). The intervention group will receive 16-weeks of education and booster sessions remotely using a video conferencing program on mini-iPads. All participants will collect a 24-hour urine specimen for sodium excretion and complete assessments of blood pressure, salt taste preference testing using salt concentration solutions, and dietary pattern using VioScreen Food Frequency Questionnaire at baseline and post intervention at 4-months. Data will be analyzed using repeated measures analysis of variance.

DETAILED DESCRIPTION:
Hypertension or high blood pressure is known as a silent killer because it can exist for decades without producing symptoms while leading to chronic cardiovascular disease and stroke. The long-term objective of this program of research is to improve blood pressure control and prevent cardiovascular disease development in adults with hypertension by increasing adherence to a sodium-restricted diet (SRD). The Sodium Watchers Program is an innovative self-management intervention using a gradual sodium adaptation strategy that allows individuals to monitor, and over time, reduce sodium content in their food, thereby increasing the ability to maintain an SRD long term. The purpose of the proposed randomized, controlled trial is to test the effects of the Sodium Watchers Program-Hypertension(SWaP-Hypertension), designed to improve blood pressure control of hypertensive adults using a gradual sodium reduction adaptation strategy.

The SWaP-Hypertension intervention consists of 14 weeks of education [4 weekly education sessions (45 minutes) followed by 5 bi-weekly sessions 5-20 minutes] that will be held at participants' preferred time delivered to their homes using a video conferencing program through a mini iPad. Using a 2-group design [SWaP-Hypertension (n=20) versus Usual care (n=10)], randomized, controlled trial with 30 hypertensive adults, the effects of the SWaP-Hypertension program on adherence to SRD, systolic and diastolic blood pressure, salt taste preference, and dietary patterns will be determined at 4 months. Data will be analyzed using repeated measures analysis of variance.

Specific Aim 1: To compare sodium intake (as reflected by 24-hour urinary sodium excretion), systolic and diastolic blood pressure, salt taste preference, and dietary patterns in the SWaP-Hypertension intervention group with the usual care group at 4 months.

Hypothesis 1: The intervention group will have a greater decline in 24-hour urinary sodium excretion and systolic and diastolic blood pressure, lower salt taste preference, and shift dietary patterns toward lower sodium foods than the usual care group at 4 months.

High blood pressure (systolic blood pressure ≥140 mmHg or diastolic blood pressure≥ 90 mm Hg), is a leading risk factor for cardiovascular disease and stroke.1 More than 80 million adult Americans have high blood pressure and it is projected that 41.4% of US adults will have hypertension by 2030.

Sodium restriction is believed to decrease blood pressure. According to a recent meta-analysis of 24 randomized controlled trials, dietary interventions (e.g., low sodium diet, low sodium/high potassium, low sodium/low calorie, Mediterranean diet, and DASH diet) were effective in reducing systolic blood pressure by an average of 3.07 mmHg and diastolic blood pressure by an average of 1.81 mmHg. These changes are minimal and are often not sustained due to the difficulty of following such diets.

Most interventions for improving adherence to SRD have focused on increasing specific skills, including how to read food labels, choose low sodium foods when eating out, and engage family support. However, these interventions do not effectively address critical barriers to SRD adherence, which include preference of high salt food and habitual dietary patterns. Salt taste reception involves the sodium ion movement through sodium channels at the apical end of the taste bud. High salt foods become preferable when individuals' taste buds adapt to foods high in sodium. Preference for salty foods results in high levels of dietary sodium intake.

These barriers are particularly salient for older patients as taste bud density decreases with age resulting in an increasing preference for salt and consumption of foods high in sodium. Combined, low palatability of low sodium foods and preference for high sodium foods make dietary changes difficult. Since at least 8-10 weeks of exposure to an SRD is required to alter sodium palatability (i.e., alter salt acuity and salt taste preference) abrupt and marked reductions in sodium intake are rarely sustained and can have the unintended consequence of exacerbating sodium-seeking behaviors. New approaches are needed to improve long-term adherence to SRD.

An innovative dietary self-care intervention has been developed to overcome sensory barriers to adherence. Abrupt and marked reductions in sodium intake can lead to sodium-seeking behaviors, and thus, changing dietary preferences requires at least 8 weeks to reach a new hedonic state and to reset sodium taste buds. Thus, an intervention that uses a gradual adaptation strategy should produce the best long-term adherence results. Most educational interventions have focused on improving knowledge by teaching patients specific skills including how to read food labels, how to choose low sodium foods when eating out, and how to modify their usual diet.

Design: A two-group, randomized, controlled design will be used to determine the effect of the SWaP-Hypertension on outcomes of hypertensive adults. A total of 30 eligible participants will be randomly assigned to intervention (n=20) or usual care group (n=10). We will assign 20 participants in the intervention that is two times more than the usual care group in order to maximize limited funding sources. The intervention will be delivered for 14 weeks using video conferencing on an iPad device. Post-intervention will be measured at 4 months follow up to examine short-term effect. Dependent variables included adherence to the SRD, systolic and diastolic blood pressure, salt taste preference, and dietary patterns.

Intervention: Sodium Watchers Program-Hypertension (SWaP-Hypertension): The SWaP- is an educational-behavioral intervention that uses an electronic salt monitoring device to promote both rural adults with high blood pressure and their family partner's ability to self-monitor sodium intake and gradually decrease their appetite for salt. The program consists of 14 weeks education [4 weekly education sessions (45 minutes) followed by 5 bi-weekly sessions (15-20 minutes)] that will be held at the dyads' preferred time delivered to their homes using a video conferencing program through a mini iPad. Video conferencing technology is used to enhance the feasibility and decrease the burden of participating in the intervention. Bi-weekly booster sessions are added to provide on-going support to maintain acquired self-care behaviors and individual goals for reductions in dietary sodium. The booster sessions include positive reinforcement of success and identification of strategies to overcome ongoing or new challenges. A nurse interventionist who experienced in delivering the intervention will assist individual goal settings and reinforces strategies in each session.

Usual care group: The usual care group receive their routine medical and nursing care for hypertension that consists of a recommendation to follow an SRD and take medications as ordered.

Measures: Table 2 lists dependent variables and their measurement in the study. To completely characterize subjects and monitor potential intervening variables, data about the individuals' age, sex, race/ethnicity, education level, comorbidities, medications, and cognitive impairment will be collected from the participant interviews or using a structured questionnaire. Comorbidity will be measured using the Charlson Comorbidity Index. Data about medications will be self-report. Cognitive impairment will be assessed using the Mini-Cog. This 3-minute screening instrument consists of drawing a clock and three-word recall. It is sensitive, reliable and valid in individuals with low literacy and low socioeconomic status. Our research staff has extensive experience in all data collection proposed in this study.

Procedure: Permission to conduct the study was obtained from the University of Kentucky, Institutional Review Board. Hypertensive adults are referred to this project by physicians and nurse practitioners from the outpatient cardiology and internal medicine services at the University of Kentucky HealthCare at Lexington. After referral, a trained research nurse will screen patients for eligibility by medical chart review. For eligible participants, the study requirements are explained and signed informed consents are obtained. After we obtain the informed consents from eligible participants, urine containers and collection devices (urinals for men and toilet "hats" for women) are provided before home visits. The participants are instructed how to collect the 24-hour urine specimen, and written standard instructions are also provided. Urine is kept in the container and does not need refrigeration. Research staff and participants set up the starting day of urine collection and pick up urine specimens in their home. During the home visit, they are assisted to complete all study questionnaires using the REDCap system and assessment of blood pressure and salt taste preference. A trained staff member will deliver education materials and an iPad to the participants in the intervention group and instruct them how to use the video conference program (i.e., Zoom Mobile app) on iPad by testing trial of a video-conferencing program. A toll-free phone number is to call at any time for assistance using the iPad is provided. The usual care group will receive a mini iPad with instruction of using emails and text message to contact research staff. All participants will follow the same data collection procedure as during the baseline assessment for 4-months follow-up time point.

ELIGIBILITY:
Inclusion Criteria:

* Systolic Blood Pressure equal to or greater than 140 mmHG and diastolic pressure equal to and greater than 90 mmHG
* Are Able to speak and write English
* Are over 40 years of age

Exclusion Criteria:

* Hypertension below the age of 40
* Major Clinical cognitive impairment
* Have major co-morbidities or co-existing terminal illnes
* Have a dietary prescription that prevents following a 2-3 gram sodium diet

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Change in oral salt taste sensitivity | up to 36 weeks
  Salt taste acuity will be tested by using the "updown" procedure. In the up trial, samples are given from lowest to highest salt concentration. Patients swish samples in the mouth for 2-3 seconds, expectorate, and then judge the saltiness of solution. The mouth is rinsed with 10 mL of distilled water between samples. When patients detect salt taste in two consecutive samples, the lower concentration of the two samples is recorded as the level of salt taste sensitivity. In the down trial, patients are given samples in reverse order from highest to lowest concentration and when no salt taste is detected in two consecutive samples, the level of salt taste sensitivity is then recorded as the concentration of the immediately preceding sample. Participants will perform this task at baseline and approximately at 20 weeks at the end of the intervention (up to 36 weeks). Data will be presented as the average as their high and low sodium sensitivity over time compared between groups.
Change in blood pressure over time | up to 36 weeks
  Systolic and diastolic blood pressures are preferred for use in hypertension classification. Mercury sphygmomanometers still are the preferred device .The position of the patient can have a sizable impact on blood pressure measurements. For the most accurate measurement, the AHA recommends that the patient be relaxed and seated with legs uncrossed and back and arm supported. For correct cuff placement, the midline of the cuff bladder should be positioned over the arterial pulsation in the patient's upper arm following palpation of the brachial artery in the antecubital fossa.The cuff should be inflated to at least 30 mm Hg above the point at which the radial pulse disappears. The cuff should then be deflated at a rate of 2 to 3 mm Hg per second. At least two readings should be taken, with a one-minute interval between them, and the average of the measurements recorded. Data will be presented as an average of the two measurements taken.
Change in adherence to sodium restricted diet over time | up to 36 weeks
  Participants will complete a 24-hour urinary sodium excretion test at baseline and at 20 weeks after the intervention is complete (up to 36 weeks). 24 hour urinary sodium excretion is tested by collecting all urine excreted over the course of 24 hours. Participants are asked to note the time when they start in a written log, then discard the first urine after that time. They will then collect all urine excreted over the course of the next 24 hours, noting down the time and amount excreted each time in the written log. Urine is stored in a container and does not need refrigeration. 24 Hour Urine Sodium Samples will be analyzed by the University of Kentucky clinical laboratory.Data will be presented as the amount of miligrams excreted per day.

SECONDARY OUTCOMES:
Change in dietary quality over time | up to 36 weeks
  Participants will complete the Vio-Food Frequency Questionnaire at baseline and 20 weeks after the intervention is complete (up to 36 weeks). This scale is a web-based food frequency questionnaire that was developed by Viocare Technologies, Inc (Princeton, NJ). It will be used to generate the Health Eating Index-20120 score which is comprised of 12 components including total fruit, whole fruit, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids, refined grains, empty calories and sodium. Each component score ranges from 0 to 100 and the high score indicates better quality of dietary component. Changes in total HEI score as well as changes in the score of each of the 12 components provide an easy, scientifically sound, quantitative way to track changes in eating patterns over time.Data will be presented as change in the Health Eating Index -2010 score over time presented as mean plus or minus standard error.
Change in Depression over time | up to 36 weeks
  Participants will complete the PHQ-9 depression scale at baseline and 20 weeks after the intervention is complete. (up to 36 weeks) This scale measures depression by answering nine questions, each question is scored on a scale of 0-3 where 0 is no depressive symptoms and 3 is considered severe depressive symptoms. A score of 1-4 is minimal depression, a score of 5-9 is mild depression, a score of 10-14 is moderate depression, a score of 15-19 is moderately severe depression, and a score of 20-27 is severe depression. Data will be presented as the change in depression over time presented as the mean plus or minus the standard error.

CONTACTS AND LOCATIONS:
Overall Officials: Misook L Chung, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time.